CLINICAL TRIAL: NCT04350931
Title: Application of BCG Vaccine for Immune-prophylaxis Among Egyptian Healthcare Workers During the Pandemic of COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Adel Khattab, Professor of chest Faculty of Medicine Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU P19a/ 2020
Record Dates: First submitted 2020-04-13; First posted 2020-04-17 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A block-randomization scheme will be generated by computer software. Participants will be randomized between 0.10 mL intradermal injection of BCG vaccine or placebo normal saline in a 2:1 ratio (600 will receive BCG & 300 will receive placebo saline). In Egypt, the available BCG vaccine is the Copenhagen (Danish strain).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG Vaccine (Active Comparator): 0.10 mL intradermal injection of BCG Vaccine over the distal insertion of the deltoid muscle onto the humerus (approximately one third down the left upper arm) slowly over 10 seconds (In Egypt, the available BCG vaccine is the Copenhagen BCG vaccine - The Danish Strain 1331 of Mycobacterium Bovis). Each 0.10 mL vaccine contains 200000-800000 colony forming units.
  Interventions: Biological: intradermal injection of BCG Vaccine
- intradermal normal saline (Placebo Comparator): placebo 0.10 mL intradermal normal saline (0.9% NaCl) over the distal insertion of the deltoid muscle onto the humerus (approximately one third down the left upper arm) slowly over 10 seconds.
  Interventions: Other: placebo

INTERVENTIONS:
Biological: intradermal injection of BCG Vaccine — 0.10 mL intradermal injection of BCG Vaccine over the distal insertion of the deltoid muscle onto the humerus (approximately one third down the left upper arm) slowly over 10 seconds
  Arms: BCG Vaccine
Other: placebo — placebo 0.10 mL intradermal normal saline (0.9% NaCl) over the distal insertion of the deltoid muscle onto the humerus
  Arms: intradermal normal saline

SUMMARY:
Phase III Placebo-controlled adaptive multi-centre randomized controlled trial Interventional (Clinical Trial). The study will include nine hundred healthcare workers in the isolation hospitals for COVID-19 cases; they will be randomly assigned to receive either BCG vaccine or normal saline.

DETAILED DESCRIPTION:
Nine hundred healthcare workers will be randomly assigned to receive intradermal injection of either BCG vaccine or normal saline.

During the study:

1. Mantoux Tuberculin skin testing (will be done prior to administration of the BCG vaccine in the first group by intradermally injecting 0.1 mL of liquid containing 5 TU (tuberculin units) of purified protein derivative (PPD) in the volar aspect of the left forearm. The test is being read after 48-72 hrs. A positive tuberculin test is defined as induration ≥10 mm.
2. Participants will be assessed clinically on daily basis for COVID 19 infection in the form of: fever, dry cough, fatigue, & dyspnea.
3. PCR sampling for COVID-19 will be withdrawn for all participants at the end of the study.
4. The duration of follow-up for each participant depends on the interim results of the primary endpoint and the probability of obtaining a result, with a maximum of 6 months.

Randomization method:

A block-randomization scheme will be generated by computer software. Participants will be randomized between 0.10 mL intradermal injection of BCG vaccine or placebo normal saline in a 2:1 ratio (600 will receive BCG & 300 will receive placebo saline). In Egypt, the available BCG vaccine is the Copenhagen (Danish strain).

End point of the study:

* Primary endpoint: Confirmed COVID-19 infection
* Secondary endpoint: number of days of (unplanned) absenteeism for any reason.
* Tertiary endpoints: number of days of (unplanned) absenteeism because of documented COVID-19 infection, and the cumulative incidence of hospital admission, ICU admission, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Healthy healthcare workers defined as nurses and physicians working at emergency rooms, ICUs, and wards of isolation hospitals

Exclusion Criteria:

* Immunosuppression
* Pregnancy & lactation
* Chronic underlying medical illness
* Known allergy to (components of) the BCG vaccine or serious adverse events to prior BCG administration
* Known active or latent Mycobacterium tuberculosis or with another mycobacterial species.
* Fever (>38 C) within the past 24 hours
* Current bacterial infection
* Recent viral infection
* Refusal of doing tuberculin test in the first group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
incidence of confirmed COVID-19 | 9 months
  Estimate the incidence of confirmed COVID-19 among the healthcare workers in isolation hospitals
Effectiveness of BCG vaccine | 9 months
  Evaluate the effectiveness of BCG vaccine in protecting the healthcare workers in isolation hospitals against the risk of COVID-19 infection by detecting any positive cases among vaccinated healthscare workers

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No